CLINICAL TRIAL: NCT00075699
Title: A Randomized Controlled Trial of Active Symptom Control With or Without Chemotherapy in the Treatment of Patients With Malignant Pleural Mesothelioma
Brief Title: Active Symptom Control With or Without Chemotherapy in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: BTS-MRC-MS01; CDR0000347461 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN54469112; EU-20349
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-06

CONDITIONS: Malignant Mesothelioma
Keywords: epithelial mesothelioma; localized malignant mesothelioma; advanced malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; Mitomycin; Vincristine; Vinorelbine; Analgesia; Psychiatric Rehabilitation

INTERVENTIONS:
Drug: cisplatin
Drug: mitomycin C
Drug: vincristine sulfate
Drug: vinorelbine tartrate
Procedure: pain therapy
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Active symptom control may decrease chest pain, breathlessness, sweating, and general discomfort in patients with malignant pleural mesothelioma. It is not yet known if active symptom control is more effective with or without chemotherapy.

PURPOSE: This randomized phase III trial is studying active symptom control and chemotherapy to see how well they work compared to active symptom control alone in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with malignant pleural mesothelioma treated with active symptom control (ASC) alone vs ASC and mitomycin, vinblastine, and cisplatin vs ASC and vinorelbine.

Secondary

* Compare the toxic effects of these regimens in these patients.
* Compare symptom palliation (chest pain, breathlessness, malaise, and sweating attacks) in patients treated with these regimens.
* Compare the performance status of patients treated with these regimens.
* Compare analgesic usage in patients treated with these regimens.
* Compare the tumor response and progression-free survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive active symptom control (ASC) through regular visits at a specialist clinic. ASC may include steroids, analgesics, appetite stimulants, bronchodilators, and/or palliative radiotherapy, when required.
* Arm II: Patients receive ASC and chemotherapy comprising mitomycin IV, vincristine IV, and cisplatin IV on day 1. Chemotherapy repeats every 21 days for a total of 4 courses.
* Arm III: Patients receive ASC and vinorelbine IV over 5 minutes weekly for 6 weeks. Vinorelbine repeats every 55 days for a total of 2 courses.

Quality of life is assessed at baseline, every 3 weeks for 21 weeks, and then every 8 weeks thereafter.

Patients are followed at 15, 18, and 21 weeks, and then every 8 weeks thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 840 patients (280 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and immunohistochemically confirmed malignant pleural mesothelioma

  * Epithelial and other histological types are allowed
  * No more than 3 months since diagnosis
* Symptomatic pleural effusion must have been treated and brought under control by drainage, pleurodesis, or pleurectomy
* Prior surgical resection of mesothelioma allowed provided 2 CT scans at least 6 weeks apart show stable or progressive disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine clearance > 50 mL/min

Pulmonary

* See Disease Characteristics

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Considered medically fit to receive chemotherapy
* No other disease or prior malignancy likely to interfere with protocol treatments or comparisons
* No clinical evidence of infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for mesothelioma

Endocrine therapy

* Not specified

Radiotherapy

* Prior local radiotherapy to a wound site after exploratory thoracotomy allowed

Surgery

* See Disease Characteristics
* See Radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2003-09

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Palliation of chest pain, breathlessness, malaise (e.g., feeling weak, tiredness, anorexia), and sweating attacks
Performance status as measured by WHO grade
Analgesic usage
Toxicity as measured by the NCIC CTC
Quality of life as assessed by the European Organization for Research and Treatment of Cancer
Tumor response as measured by the RECIST criteria
Progression-free survival as measured by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Martin F. Muers, MD, Principal Investigator — Leeds General Infirmary
Locations (3):
- United Kingdom (3):
  - Leeds General Infirmary at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England

REFERENCES:
- [Background] Muers MF, Rudd RM, O'Brien ME, Qian W, Hodson A, Parmar MK, Girling DJ; British Thoracic Society Mesothelioma Group. BTS randomised feasibility study of active symptom control with or without chemotherapy in malignant pleural mesothelioma: ISRCTN 54469112. Thorax. 2004 Feb;59(2):144-8. doi: 10.1136/thorax.2003.009290. PMID 14760156
- [Background] Qian W, Muers MF, Rudd RM, et al.: A feasibility study of active symptom control (ASC) with or without chemotherapy in malignant pleural mesothelioma. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2568, 639, 2003.
- [Result] Muers MF, Stephens RJ, Fisher P, Darlison L, Higgs CM, Lowry E, Nicholson AG, O'Brien M, Peake M, Rudd R, Snee M, Steele J, Girling DJ, Nankivell M, Pugh C, Parmar MK; MS01 Trial Management Group. Active symptom control with or without chemotherapy in the treatment of patients with malignant pleural mesothelioma (MS01): a multicentre randomised trial. Lancet. 2008 May 17;371(9625):1685-94. doi: 10.1016/S0140-6736(08)60727-8. PMID 18486741
- [Result] Muers M, Fisher P, Snee M, et al.: A randomized phase III trial of active symptom control (ASC) with or without chemotherapy in the treatment of patients with malignant pleural mesothelioma: first results of the Medical Research Council (MRC) / British Thoracic Society (BTS) MS01 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA7525, 390s, 2007.